CLINICAL TRIAL: NCT03458221
Title: Signal TrAnsduction Pathway Activity Analysis in OVarian cancER
Acronym: STAPOVER
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gynaecologisch Oncologisch Centrum Zuid (Other)
Collaborators: Radboud University Medical Center (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); InnoSIGN (Unknown); Eurofins (Industry)
Responsible Party: Principal Investigator, Jurgen M.J. Piek, MD, PhD, Catharina Ziekenhuis Eindhoven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAPOVER; 2020-005091-36 (EudraCT Number)
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Recurrent Ovarian Cancer; Signal Transduction Pathway Deregulation; Therapy-Associated Cancer
Keywords: Ovarian Cancer; Signal Transduction Pathway; Targeted therapy; Drug repurposing
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Intervention Model Description: Targeted therapy based on functional signal transduction pathway activation in patients with recurrent ovarian cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A - ER active tumors (Experimental): In case of an aberrantly active Estrogen Receptor (ER) pathway, patients will be treated with Letrozole 2.5mg daily orally until progression of disease.
  Interventions: Drug: Letrozole Oral Product
- B - AR active tumors (Experimental): In case of an aberrantly active androgen receptor (AR) pathway, patients will be treated with Bicalutamide 150mg daily orally until progression of disease.
  Interventions: Drug: Bicalutamide Oral Product
- C - PI3K active tumors (Experimental): In case of an aberrantly active phosphoinositide 3-kinase (PI3K) pathway, patients will be treated with Everolimus 10mg daily orally until progression of disease.
  Interventions: Drug: Everolimus Oral Product
- D - HH and/or PI3K active tumors (Experimental): In case of an aberrantly active Hedgehog (HH) or PI3K pathway, patients will be treated with Itraconazole 300mg twice daily orally until progression of disease.
  Interventions: Drug: Itraconazole Oral Product

INTERVENTIONS:
Drug: Letrozole Oral Product — Letrozole 2.5mg tablet - 2.5mg once dailty until progression of disease.
  Arms: A - ER active tumors
Drug: Bicalutamide Oral Product — Bicalutatmide 150mg tablet - 150mg once daily until progression of disease.
  Arms: B - AR active tumors
Drug: Everolimus Oral Product — Everolimus 10mg tablet - 10mg once daily until progression of disease.
  Arms: C - PI3K active tumors
Drug: Itraconazole Oral Product — Itraconazole 100mg capsule - 300mg twice daily until progression of disease.
  Arms: D - HH and/or PI3K active tumors

SUMMARY:
The purpose of this prospective, parallel-group, cohort study is to implement phenotype-guided targeted therapy based on functional signal transduction pathway (STP) activity in recurrent ovarian cancer patients using a novel mRNA-based assay. Existing targeted drugs with tolerable toxicity profiles are used to investigate the therapeutic value beyond their approved indication, which are deemed beneficial in the select group of patients with a relevant predominantly active functional STP, in order to improve survival and maintain quality of life.

DETAILED DESCRIPTION:
Rationale: Ovarian cancer is one of the most lethal cancers in the world. Standard therapy consists of debulking surgery and chemotherapy. However, despite this aggressive treatment, recurrent disease almost invariably occurs resulting in a five-year survival rate of approximately 30%. Tumour growth is driven by several signal transduction pathways (STPs), and twelve major STPs have been identified as important for carcinogenesis. Currently, several targeted therapy drugs are available and new targeted drugs are being developed. With a newly developed technique, Signal Transduction Activation (STA) analysis, it is possible to assess which pathway is predominant in a specific (ovarian) cancer sample. Therefore, we hypothesize that specifically targeting the predominant STP might impair tumour growth and improve survival.

Objective: This study aims to investigate the progression-free survival (PFS) according to RECIST 1.1 criteria on matched targeted therapy by STA-analysis (PFS2) in comparison to the PFS recorded on the therapy administered immediately prior to enrolment (PFS1) in women with recurrent ovarian cancer.

Study design: A multi-centre prospective, parallel-group, cohort study. Study population: Recurrent ovarian cancer patients with platinum-resistant disease, patients who refrain from standard therapy and patients who are not yet eligible for standard palliative chemotherapy, including all histological subtypes.

Intervention: STA-analysis will be performed on a biopsy taken from the recurrent tumour. Patients will be included if a predominant pathway is identified for which a matched targeted drug is available and deemed adequate by the multidisciplinary tumour board. We will start with targeted therapy in patients with oestrogen receptor, androgen receptor, phosphoinositide 3-kinase and Hedgehog pathway active tumours, since targeted therapy interceding these pathways are easily available with tolerable side effects.

Main study parameters/endpoints: The primary outcome is therapy response defined as PFS2/PFS1 ratio according to RECIST 1.1 criteria. Secondary outcomes include the proportion of patients with an actionable active pathway and the proportion of patients receiving matched targeted therapy, best overall response (according to RECIST 1.1 criteria), one-year survival, overall survival, predictive value of STA-analysis results, side effects, quality of life, cost-effectiveness and change in STP activity score comparing the score before treatment and after disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Female, age > 18 years
* Patients with recurrent ovarian cancer who meet one of the following criteria:
* Platinum-resistant disease, defined as disease recurrence or progression within six months of last platinum-based chemotherapy or;
* Patient refrains from standard therapy or;
* Asymptomatic patient who is not yet eligible for standard palliative chemotherapy but has an increase of CA125 tumour marker at two consecutive time points 28 days apart with a value of two times nadir above 35 U/ml.
* Progressive disease after at least one prior line of systemic treatment for recurrent disease.
* Radiologically evaluable disease according to RECIST 1.1 criteria (36).
* Ability and willingness to obtain a tumour biopsy after the last course of standard treatment and before start of the study.
* Ability and willingness to provide written and oral consent.
* Able to speak and understand the Dutch language.
* WHO performance status 0-II.
* Adequate renal and liver function to start matched targeted therapy (according to the local clinician).
* Adequate use of contraceptives in case of patients with childbearing potential.

Exclusion Criteria:

* Age < 18 years.
* Patient is receiving any other anti-cancer therapy (e.g. cytotoxic or targeted drug or radiation) or is chemotherapy naïve. The required wash out period prior to start of matched targeted therapy is at least three weeks.
* Patient is diagnosed with or treated for a second primary tumour (except non-melanoma skin tumour) one year prior to study inclusion.
* Inability to obtain (sufficient) tumour material.
* Previous use of the selected targeted drug as anti-cancer agent.
* Physical condition WHO III-IV.
* Pregnant or lactating women.
* Simultaneous participation in another treatment-related clinical trial.
* Patients with any other clinically significant medical condition which, in the opinion of the local clinician, makes it undesirable for the patient to participate in this study or which could jeopardize compliance with study requirements including, but not limited to: ongoing or active infection, severe psychiatric illness, or complicated social situations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer
Enrollment: 148 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival on matched targeted therapy determined by STP-activity (PFS2) in comparison to the PFS recorded on the therapy administered immediately prior to enrolment (PFS1). | From baseline until the date of documented disease progression or 12 months after the start of targeted therapy.
  PFS on matched targeted therapy (PFS2) is defined as the time from start of matched targeted therapy to disease progression, defined by RECIST 1.1 criteria, or death from any cause. PFS on prior therapy (PFS1) is defined as the time from start of the prior treatment to disease progression defined by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Proportion of patients with an actionable active pathway for which targeted therapy is recommended in relation to the number of patients who underwent a biopsy. | From date of biopsy until the date of the result from Multi-disciplinary Tumor Board Meeting, up 14 days after biopsy date.
Proportion of patients who receive matched targeted therapy in relation to the number of patients included in each study arm. | From start date matched targeted therapy until the end of the study enrollment, up to 36 months.
  Proportion of patients included in arm A, B, C, D.
Best overall response defined by RECIST 1.1 criteria based on radiological imaging. | From baseline, radiological evaluation every 12 weeks after the start of targeted therapy until the date of documented disease progression or death, whichever comes first, assessed up to 12 months.
One-year survival | From start date of targeted therapy until date of death or one year follow-up, whichever comes first.
  One-year survival is defined as the time from start matched targeted therapy till death or the end of the one-year follow-up period.
Overall survival | From start date of targeted therapy until the date of death, assessed up to 36 months.
  Defined as the time from start matched targeted therapy till death.
Predictive value of STA-analysis results on matched targeted therapy response. | From start date targeted therapy until response evaluation at 12 weeks after start of targeted therapy.
Side effects | From start date of targeted therapy after two weeks, every 12 weeks from targeted therapy start date, until 12 weeks after end of treatment.
  Assessed according to the PRO-CTCAE and NCI CTCAE 5.0
Health Related Quality of Life | From baseline, every 12 weeks after start date of treatment until 12 weeks after end of treatment.
  HRQoL is assessed using standardized questionnaires from the EORTC QLQ-C30 and QLQ-OV28.
Cost-effectiveness | From baseline, every 12 weeks after start date of targeted therapy until 12 weeks after end of treatment.
  Standardized EuroQol 5D (EQ-5D-5L) questionnaire is used to calculated the cost-effectiveness.
Change in pathway activity score after disease progression compared to pathway activity score before start of matched therapy. | From date of biopsy until 4 weeks after date of documented progression of disease.
  If pathway activity scores are available from a second (voluntary) biopsy for after treatment has ended and before standard (palliative) treatment has started, change in pathway scores are assessed.

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Radboudumc, Nijmegen, Gelderland
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Amphia Hospital, Breda
  - Maastricht UMC+, Maastricht
  - Erasmus MC, Rotterdam
  - Elisabeth-Tweesteden Hospital, Tilburg

IPD SHARING:
Plan to Share IPD: Undecided